CLINICAL TRIAL: NCT00634920
Title: A Controlled Randomized Open-label Multicenter Study Evaluating if Early Conversion to Everolimus (Certican) From Cyclosporine (Neoral) in de Novo Renal Transplant Recipients Can Improve Long-term Renal Function and Slow Down the Progression of Chronic Allograft Nephropathy
Brief Title: Evaluation of Early Conversion to Everolimus From Cyclosporine in de Novo Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ASE01; 2007-000771-42 (EudraCT Number)
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Renal Function
Keywords: De novo renal transplantation
MeSH Terms: interventions — Everolimus; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones; Prednisolone; Basiliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (CNI-free) (Experimental): Patients in this group were converted to everolimus immunosuppressive therapy. The patients in the everolimus group were treated with everolimus, off-label (CNI-free) use, and EC-MPS and corticosteroids in accordance with local practice and approved label. Conversion to everolimus was as follows: Day 1: begin everolimus 3 mg in the evening. Usual morning dose of CsA and 50% reduced evening dose of CsA Day 2: everolimus 2 mg in the morning and 2 mg in the evening, complete discontinuation of CsA Day 3 or 4, and onwards: everolimus according to trough level 6-10 ng/mL.The given total daily dose of the immunosuppressive drugs (everolimus) was divided into two (equal) doses, applied 12 hours apart.
  Interventions: Drug: everolimus; Drug: Enteric Coated Mycophenolate Sodium (EC-MPS); Drug: corticosteroids; Drug: Basiliximab
- Control (CsA) (Active Comparator): Patients in the control group continued on an immunosuppressive regimen. The patients in this Control group were treated with CsA, EC-MPS and corticosteroids in accordance with local practice and approved label. The given total daily dose of the immunosuppressive drugs (CsA and EC-MPS) was divided into two (equal) doses, applied 12 hours apart.
  Interventions: Drug: cyclosporine A; Drug: Enteric Coated Mycophenolate Sodium (EC-MPS); Drug: corticosteroids; Drug: Basiliximab

INTERVENTIONS:
Drug: everolimus — Everolimus (Certican®) tablets administered orally in two divided doses (b.i.d.) at a starting dose of 4 mg/day adjusted to target a trough blood concentration between 6 and 10 ng/mL in period 2.
  Other Names: Certican
  Arms: Everolimus (CNI-free)
Drug: cyclosporine A — CsA (Sandimmun Neoral), based on C0-h levels 75-200 ng/mL or C2-h levels 700 900 ng/mL from randomization to Month 6, or C0-h levels 50-150 ng/mL or C2-h levels 600 800 ng/mL from Month 6 to Month 36, according to local method
  Other Names: Sndimmun Neoral
  Arms: Control (CsA)
Drug: Enteric Coated Mycophenolate Sodium (EC-MPS) — Target dose 1440 mg in the control group, target dose 1080 in the everolimus group (higher dose in the CsA group because of interactions of CsA on gastric reabsorption of mycophenolate)
  Other Names: Myfortic
Drug: corticosteroids — For both groups: minimum corticosteroid dose of 10 mg until week 12, 5-10 mg until month 12, month 12-36 corticosteroid treatment on investigator's descretion.
  Other Names: Prednisolone
Drug: Basiliximab — Induction therapy 20 mg basiliximab on Day 0 prior to reperfusion and 20 mg on Day 4 post-TX.
  Other Names: Simulect

SUMMARY:
This study is designed to evaluate if early conversion to everolimus from cyclosporine in de novo renal transplant recipients can improve long-term renal function and slow down the progression of chronic allograft nephropathy

ELIGIBILITY:
Inclusion Criteria:

* First or second single renal transplant from deceased or living donor

Exclusion criteria

* Recipient of organs other than a renal transplant
* Present malignancy (within the last 2 years) other than excised basal cell or squamous cell carcinoma of the skin
* Severe liver disease
* At the time of randomization 7 weeks after transplantation

In addition to the above criteria the following must be met at time of randomization:

Inclusion Criteria:

* Patients maintained on a triple immunosuppressive regime consisting of cyclosporine, Enteric coated mycophenolate, and corticosteroids
* Patients completed the first 7 weeks without experiencing any rejection

Exclusion Criteria:

* Graft loss
* Low hemoglobin value, low number of white blood cells or platelets
* High cholesterol values
* Proteinuria
* Wound healing problems
* Current severe major local or systemic infection
* Renal insufficiency

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Denmark (4):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense C
- Novartis Investigative Site, Oslo, Norway
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Uppsala

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 periods, period 1: TX to Week 7 ± 7 days post-TX and period 2: Week 7 ± 7 days post-TX to Month 36. 341 patients were enrolled in this study. 204 randomized to receive study treatment: 104 in the everolimus group, 100 in the control group. 2 patients in everolimus group did not receive at least one dose of study treatment.
Groups:
- Everolimus (CNI-free): This investigational drug was provided by Novartis. All patients received induction therapy with basiliximab, and commenced on an immunosuppressive regimen consisting of CsA, EC-MPS and corticosteroids before they were randomized. After randomization patients in the everolimus group (CNI-free regimen) were treated with everolimus (Certican) EC MPS and corticosteroids. Patients randomized to this arm 7 weeks after renal transplantation will do an overnight switch from cyclosporine to everolimus.
- Control (CsA): All patients received induction therapy with basiliximab, and commenced on an immunosuppressive regimen consisting of CsA, EC-MPS and corticosteroids before they were randomized. After randomization patients in the control group continued on the prior immunosuppressive regimen given before randomization. Conventional treatment arm with cyclosporine (CsA), mycophenolate (Myfortic) and corticosteroids continued for the entire 36 months study period.
- Pre-Randomized Patients: All patients received induction therapy with 20 mg basiliximab on Day 0 prior to reperfusion and 20 mg at Day 4 post-TX (transplatation), and commenced on an immunosuppressive regimen consisting of: CsA (based on trough levels C0-h 100-250 ng/mL or C2-h 900 1300 ng/mL, according to local method), EC MPS (target dose 1440 mg/day, minimum dose 1080 mg/day at the time of randomization), Corticosteroids (a minimum dose of 10 mg prednisolone or equivalent was given at time of randomization).
Period: Period 1 - Pre-Randomization
Arm/Group | Everolimus (CNI-free) | Control (CsA) | Pre-Randomized Patients
Started | 0 | 0 | 341 (Total number of Enrolled patients)
Completed | 0 | 0 | 204 (Total number of patients who became randomized)
Not Completed | 0 | 0 | 137
Not completed — Adverse Event | 0 | 0 | 36
Not completed — Wound healing problems | 0 | 0 | 16
Not completed — Rejections | 0 | 0 | 55
Not completed — Withdrawal by Subject | 0 | 0 | 21
Not completed — Non-Compliance | 0 | 0 | 3
Not completed — Other issues | 0 | 0 | 6
Period: Period 2 - Post-Randomization
Arm/Group | Everolimus (CNI-free) | Control (CsA) | Pre-Randomized Patients
Started | 104 (2 patients randomized in this group did not receive at least one dose of study drug.) | 100 | 0 (This group included patients who had renal TX but did not qualify for randomization at Visit 2.)
Full Analysis Set (FAS) | 92 | 90 | 0
Completed | 43 | 68 | 0
Not Completed | 61 | 32 | 0
Not completed — Adverse Event | 37 | 9 | 0
Not completed — Rejection | 11 | 5 | 0
Not completed — Death | 2 | 5 | 0
Not completed — consent withdrawal, non compliance | 9 | 13 | 0
Not completed — Patients did not receive study drug | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized Patients: This group included patients in whom a renal TX was performed but who did not qualify for randomization at Visit 2. This group was to be described with respect to treatment, reason for not randomized and outcome variables calculated or measured GFR, whichever was feasible, BPAR, graft loss or death at 12 months (no outcome variables were collected for this population
- Total: Total of all reporting groups
Arm/Group | Everolimus (CNI-free) | Control (CsA) | Not Randomized Patients | Total
Number analyzed (Participants) | 104 | 100 | 137 | 341
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (10.9) | 53.3 (12.3) | 56.3 (12.5) | 55.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 26 | 43 | 103
  Male | 70 | 74 | 94 | 238
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 101 | 100 | 136 | 337
  Black | 1 | 0 | 0 | 1
  Oriental | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Measured Glomerular Filtration Rate
Description: To compare the efficacy between treatment regimens by assessing the difference in renal function evaluated by mean measured glomerular filtration rate (mGFR) 12 months after renal transplantation (TX). The mGFR was measured using Iohexol or Cr-EDTA clearance according to local practice.
Time Frame: Month 12
Population: The full analysis set (FAS) population consists of all randomized patients who received at least one dose of any immunosuppressive therapy after TX and have both baseline and Month 12 assessment of the primary efficacy variable (renal function based on mGFR).
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
mL/min/1.73m^2 | 51.5 (14.4) | 47.8 (15.4)

2. Secondary Outcome: Measured Glomerular Filtration Rate
Description: Progression of renal function measured by mean mGFR at 36 months after renal TX. The mGFR was measured using Iohexol or Cr-EDTA clearance according to local practice.
Time Frame: Month 36
Population: The full analysis set (FAS) population consists of all randomized patients who received at least one dose of any immunosuppressive therapy after TX and have both baseline and Month 12 assessment of the primary efficacy variable (renal function based on mGFR). Patients who did not provide mGFR assessment at M36 visit were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 87 | 90
mL/min/1.73m^2 | 48.2 (14.7) | 46.1 (17.0)

3. Secondary Outcome: Calculated Glomerular Filtration Rate
Description: The GFR was calculated according to the Modification of Diet in Renal Disease Study Group (MDRD) method, the Cockcroft-Gault method, and the Nankivell formula. cGFR was calculated from blood samples collected at predefined time points.
Time Frame: Months 12, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
mL/min/1.73m^2
  MDRD M12 | 65.0 (19.9) | 60.1 (19.7)
  MDRD M36 | 59.4 (20.1) | 57.4 (20.2)
  Cockcroft-Gault M12 | 45.4 (14.6) | 45.6 (15.4)
  Cockcroft-Gault M36 | 43.1 (16.1) | 42.1 (13.1)
  Nankivel M12 | 66.3 (19.2) | 61.8 (20.5)
  Nankivel M36 | 61.8 (20.9) | 58.9 (20.0)

4. Secondary Outcome: Progression of Measured Glomerular Filtration Rate
Description: Change in renal progression measured by mean mGFR from week 7 to Month 36
Time Frame: Week 7, Week 52, Month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
mL/min/1.73m^2
  Week 7 | 46.3 (13.0) | 47.8 (15.0)
  Week 52 | 51.5 (14.4) | 47.8 (15.4)
  Change from week 7 to Week 52 | 5.6 (11.5) | 0.0 (12.9)
  Month 36 | 48.2 (14.7) | 46.1 (17.0)
  Change from week 7 to Month 36 | 1.3 (14.0) | -1.7 (15.4)

5. Secondary Outcome: Percentage of Participants Who Developed CAN (Chronic Allograft Nephropathy)
Description: Assessed by protocol biopsies findings (Banff 1997 lesion scores and morphometry of the interstitial space)
Time Frame: Month 12, Month 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  Month 12 | 1.0 | 1.0
  Month 36 | 59.0 | 64.0

6. Secondary Outcome: Percentage of Participants With Biopsy Proven Acute Rejection (BPAR)
Description: A BPAR was defined as a biopsy graded IA, IB, IIA, IIB, or III (Banff 97 classification). Biopsy graded IA: Significant interstitial infiltration (> 25% of parenchyma) and foci of moderate tubulitis (> 4 mononuclear cells/tubular cross section or group of 10 tubular cells). Biopsy grade IB: Significant interstitial infiltration (> 25% of parenchyma) and foci of severe tubulitis (> 10 mononuclear cells/tubular cross section or group of 10 tubular cells). Biopsy grade IIA: Mild to moderate intimal arteritis. Biopsy graded IIB: Severe intimal arteritis comprising > 25% of the lumenal area.
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  Month 12: lA | 19.6 | 4.4
  Month 12: lB | 10.9 | 0.0
  Month 12: llA | 2.2 | 2.2
  Month 12: llB | 2.2 | 1.1
  Month 24: lA | 5.4 | 4.4
  Month 24: lB | 1.1 | 3.3
  Month 36: lA | 2.2 | 1.1
  Month 36: lB | 1.1 | 0.0

7. Secondary Outcome: Percentage of Participants With Graft Loss or Death
Description: The allograft was presumed to be lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis. If the patient underwent a graft nephrectomy, the day of nephrectomy was the day of graft loss. Graft loss was considered an SAE (serious adverse event).
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  Month 12: Event First Year | 0.0 | 0.0
  Month 12: No Event First Year | 100.0 | 100.0
  Month 24: Event Second Year | 1.1 | 1.1
  Month 24: No Event Second Year | 98.9 | 98.9
  Month 36: Event Third Year | 0.0 | 2.2
  Month 36: No Event Third Year | 100.0 | 97.8

8. Secondary Outcome: Time to Treatment Failure
Description: Treatment failure was defined as graft loss or death.Time to treatment failure is shown as mean time to treatment failure.
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Days | 972.7 (7.76) | 959.5 (7.76)

9. Secondary Outcome: Percentage of Participants With Treatment Failures
Description: Treatment failure was defined as graft loss or death.
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  Month 12: No Failure | 100.0 | 100.0
  Month 12: Failure | 0.0 | 0.0
  Month 24: No Failure | 98.8 | 98.8
  Month 24: Failure | 1.2 | 1.2
  Month 36: No Failure | 98.8 | 96.7
  Month 36: Failure | 1.2 | 3.3

10. Secondary Outcome: Time to First Malignancy
Description: This is the time to first diagnosed malignancy. Malignancies (skin- or solid cancer) were listed whether they reoccurred in situ, were metastatic or de novo. This is shown as mean time.
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Months
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Months | 35.5 (0.63) | 35.1 (0.55)

11. Secondary Outcome: Lipid Profile for Apolipoprotein
Description: Blood lipid levels of patients in both groups for Apolipoprotein (Apo) A1 and B.
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
g/L
  Month 12: Apolipoprotein A1 | 1.59 (0.31) | 1.46 (0.26)
  Month 24: Apolipoprotein A1 | 1.55 (0.29) | 1.36 (0.06)
  Month 36: Apolipoprotein A1 | 1.70 (0.39) | 1.56 (0.33)
  Month 12: Apolipoprotein B | 0.935 (0.235) | 0.923 (0.258)
  Month 24: Apolipoprotein B ( | 1.178 (0.225) | 1.058 (0.263)
  Month 36: Apolipoprotein B | 0.984 (0.211) | 0.934 (0.206)

12. Secondary Outcome: Lipid Profile for HDL-C, LDL-C,Total Cholesterol, and Triglycerides
Description: Blood lipid levels of patients in both groups: HDL-C, LDL-C,Total cholesterol, and triglycerides.
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
mmol/L
  Month 12: HDL Cholesterol | 1.486 (0.446) | 1.419 (0.409)
  Month 24: HDL Cholesterol | 1.477 (0.437) | 1.409 (0.411)
  Month 36: HDL Cholesterol | 1.495 (0.440) | 1.529 (0.518)
  Month 12: LDL Cholesterol | 3.569 (1.390) | 3.130 (0.962)
  Month 24: LDL Cholesterol | 3.381 (1.139) | 2.925 (1.043)
  Month 36: LDL Cholesterol | 3.206 (0.945) | 2.822 (0.789)
  Month 12: Total Cholesterol | 6.091 (1.650) | 5.318 (1.067)
  Month 24: Total Cholesterol | 5.823 (1.377) | 5.112 (1.096)
  Month 36: Total Cholesterol | 5.595 (1.396) | 4.830 (1.166)
  Month 12: Triglycerides | 2.461 (1.620) | 1.868 (0.932)
  Month 24: Triglycerides | 2.288 (1.400) | 1.757 (0.958)
  Month 36: Triglycerides | 2.164 (1.256) | 1.580 (0.853)

13. Secondary Outcome: Number of Lipid-lowering Drugs Taken
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of lipid-lowering drugs
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Number of lipid-lowering drugs
  Month 12 | 0.9 (0.4) | 0.8 (0.4)
  Month 24 | 1.0 (0.4) | 0.9 (0.4)
  Month 36 | 0.9 (0.5) | 0.8 (0.4)

14. Secondary Outcome: Percentage of Participants on Lipid-lowering Drugs
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  Month 12 | 75.0 (0.4) | 60.0 (0.4)
  Month 24 | 78.0 (0.4) | 65.0 (0.4)
  Month 36 | 73.0 (0.5) | 63.0 (0.4)

15. Secondary Outcome: Number of Antihypertensive Drugs Taken
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of antihypertensive dugs
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Number of antihypertensive dugs
  Month 12 | 2.5 (1.4) | 2.5 (1.1)
  Month 24 | 2.5 (1.3) | 2.4 (1.1)
  Month 36 | 2.0 (1.4) | 2.2 (1.3)

16. Secondary Outcome: Percentage of Participants on Antihypertensive Drugs
Time Frame: Months 12, 24, 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  Month 12: No antihypertensive drugs | 9.2 | 3.3
  Month 12: Has antihypertensive drugs | 90.8 | 96.7
  Month 24: No antihypertensive drugs | 4.2 | 5.3
  Month 24: Has antihypertensive drugs | 95.8 | 94.7
  Month 36: No antihypertensive drugs | 15.6 | 12.8
  Month 36: Has antihypertensive drugs | 84.4 | 87.2

17. Secondary Outcome: Proteinuria (Measured as Urine Albumin/Creatinine Ratio (mg/mmol))
Description: Proteinuria is when a large amount of protein, that should remain circulating in a person's blood, is "spilled" into their urine and eliminated from the body.
Time Frame: Months 12, 24, 36
Population: The safety population (SAF) consists of all patients in whom TX was performed and who were randomized and treated with at least one dose of randomized treatment.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 102 | 100
mg/mmol
  Month 12 | 17.31 (29.39) | 11.27 (22.92)
  Month 24 | 62.83 (178.62) | 24.55 (52.07)
  Month 36 | 78.78 (357.45) | 80.73 (534.30)

18. Secondary Outcome: Percentage of Participants Who Had Donor Specific Antibodies (DSA)
Description: Venous blood was drawn for donor specific (DSA) measurements prior to transplantation and at the final visit (36 months). The blood sample was first screened for the presence of PRA i.e. donor specific Immunoglobulin-G antibodies against specific HLA antigens. If PRA antibodies were detected, the blood sample was tested for specific DSAs on single antigen Luminex beads (coated with single HLA class I or II molecules). In this way, the specificity of these antibodies could be determined.
Time Frame: Month 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
Percentage of participants
  ND (not done) | 7.0 | 9.0
  Negative | 78.0 | 70.0
  Positive | 15.0 | 21.0

19. Secondary Outcome: Health-related Quality of Life (QoL) as Measured by EuroQoL EQ-5D
Description: Health-related QoL was assessed using the EQ-5D questionnaire. The EQ-5D self-report questionnaire consists of the EQ-5D descriptive system that measures health-related quality of life on 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which can take one of three responses. The responses record three levels of severity (no problems/moderate problems/severe problems) within a particular EQ-5D dimension. Scores are transformed to a range of 0-1, in which higher scores reflect better health status.
Time Frame: Before randomization, Months 12, 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Everolimus (CNI-free) | Control (CsA)
Number analyzed (Participants) | 92 | 90
scores on a scale
  Before Randomization (Week 7) | 0.8430 (0.1539) | 0.8693 (0.1583)
  Month 12 | 0.8155 (0.1605) | 0.8470 (0.2239)
  Month 36 | 0.8285 (0.2303) | 0.8422 (0.1941)

ADVERSE EVENTS:
Arm/Group | Control (CsA) | Everolimus (CNI-free)
Serious Adverse Events (participants affected / at risk) | 65/100 | 72/102
Other Adverse Events (participants affected / at risk) | 88/100 | 93/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (CsA) (N=100) | Everolimus (CNI-free) (N=102)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Polycystic liver disease (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 2 | 4
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 3
Metaplasia (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 7
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Graft versus host disease (Immune system disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 9 | 4
Abscess (Infections and infestations) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Campylobacter infection (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 1
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 6 | 4
Device related infection (Infections and infestations) | 0 | 1
Epstein-Barr viraemia (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 8
Gastroenteritis caliciviral (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2
Infected lymphocele (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 1 | 4
Lung infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 6 | 15
Pyelonephritis (Infections and infestations) | 5 | 4
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 5
Subcutaneous abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 10 | 10
Urosepsis (Infections and infestations) | 3 | 4
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 4
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0
Blood creatinine increased (Investigations) | 4 | 8
Norovirus test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 2
Monoparesis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 3
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 2
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Manual lymphatic drainage (Surgical and medical procedures) | 1 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Vesicoureteral reflux surgery (Surgical and medical procedures) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 3 | 4
Thrombosis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (CsA) (N=100) | Everolimus (CNI-free) (N=102)
Anaemia (Blood and lymphatic system disorders) | 12 | 24
Leukopenia (Blood and lymphatic system disorders) | 10 | 15
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 14
Diarrhoea (Gastrointestinal disorders) | 15 | 12
Gingival hyperplasia (Gastrointestinal disorders) | 10 | 0
Fatigue (General disorders) | 8 | 3
Oedema (General disorders) | 4 | 13
Oedema peripheral (General disorders) | 28 | 32
Cytomegalovirus infection (Infections and infestations) | 8 | 5
Gastroenteritis (Infections and infestations) | 6 | 6
Herpes zoster (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 21 | 16
Oral fungal infection (Infections and infestations) | 1 | 6
Pneumonia (Infections and infestations) | 6 | 9
Upper respiratory tract infection (Infections and infestations) | 7 | 6
Urinary tract infection (Infections and infestations) | 31 | 30
Wound (Injury, poisoning and procedural complications) | 2 | 6
Blood creatinine increased (Investigations) | 13 | 5
Polyomavirus test positive (Investigations) | 9 | 10
Gout (Metabolism and nutrition disorders) | 11 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 12 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 10
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Dizziness (Nervous system disorders) | 8 | 1
Headache (Nervous system disorders) | 6 | 8
Depression (Psychiatric disorders) | 8 | 3
Proteinuria (Renal and urinary disorders) | 4 | 14
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Acne (Skin and subcutaneous tissue disorders) | 2 | 14
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 8 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 10
Lymphocele (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.